CLINICAL TRIAL: NCT07215884
Title: Dopamine and Sensorimotor Function in Stuttering
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1R21DC021557-01A1 (NIH); R21DC021557 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Stuttering, Adult
Keywords: Stuttering; Aripiprazole; Adults with Stuttering; Speech Fluency; Auditory Feedback
MeSH Terms: conditions — Stuttering | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single dose of aripiprazole (Active Comparator): Single dose of aripiprazole, 10mg administered orally. Participant and administrator will be blinded.
  Interventions: Drug: Aripiprazole 10 MG
- Placebo dose (Placebo Comparator): A single placebo dose will be administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole 10 MG — The effects of aripiprazole on stuttering and various behavioral and neural outcomes will be studied compared to placebo.
  Arms: Single dose of aripiprazole
Drug: Placebo — Placebo will be compared against aripiprazole for effect on stuttering and various behavioral and neural markers.
  Arms: Placebo dose

SUMMARY:
This study is being done to understand the effect of aripiprazole on adults who stutter. Stuttering is a disorder that affects speech fluency. This study aims to understand sensorimotor pathways of stuttering and possible interventions.

DETAILED DESCRIPTION:
Stuttering is a disorder of speech fluency that affects 3.5 million people in the USA alone. The goal of this project is to assess whether fluency ehnancement with auditory feedback manipulations or with pharmacological agents that regulate dopamine uptake improve the sensorimotor functions of speech feedback prediction and processing in stuttering.

This study may lay the foundation for stuttering treatments that combine dopamine regulators and behavioral treatments. Aripiprazole is an FDA-approved anti-psychotic typically used for treatment of schizophrenia or acute manic episodes. A typical dose is 10-15 mg per day, given daily for treatment. In this study, one 10 mg dose will be given. The usage in this study is purely investigational (experimental) and not FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* native speakers of American English
* for adults who stutter, presence of stuttering will be confirmed, with onset before age 6 years
* Normal hearing
* Ages of 18 to 65 years
* healthy adults without hearing-language difficulties

Exclusion Criteria:

* self-reported speech-language-hearing difficulties other than stuttering
* self-reported neurological or psychological problems
* other medications (drugs that affect dopaminergic system and/or benzodiazepines)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pre-speech auditory modulation | 3-4 hours after intervention dose is delivered
  Pre-speech auditory modulation (PSAM) is a measure of auditory cortical activity (as collect via magnetoencephalography) in response to a speaking and and matching silent reading task.
Speaking Induced Suppression (SIS) | 3-4 hours after intervention
  SIS is a phenomenon measured through magnetoencephalography that is a marker of auditory cortical response to self-produced speech compared with playback of the same speech.
Centering | 3-4 hours after intervention
  This is a speech behavior associated with SIS involving a reduction of speech variability from speech onset to mid-utterances. This is derived from auditory recordings occurring during magnetoencephalography collection.
Feedback alterations | 3-4 hours after intervention
  This is a measure of fluency enhancement by altered speech feedback (manipulated by methods such as masking noise, frequency shifted feedback,. etc.) This is measured through audio recordings and brain activation patterns during magnetoencephalography.

CONTACTS AND LOCATIONS:
Overall Officials: John Houde, PhD, Principal Investigator — University of California, San Francisco; Srikantan Nagarajan, PhD, Principal Investigator — University of California, San Francisco; Ludo Max, PhD, Principal Investigator — University of Washington
Locations (1):
- Biomagentic Imaging Lab, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Audio and video recordings to verify presence of stuttering will be shared with investigators at University of Washington. De-identified MEG data or results may also be shared with University of Washingotn.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Toyomura A, Miyashiro D, Kuriki S, Sowman PF. Speech-Induced Suppression for Delayed Auditory Feedback in Adults Who Do and Do Not Stutter. Front Hum Neurosci. 2020 Apr 24;14:150. doi: 10.3389/fnhum.2020.00150. eCollection 2020. PMID 32390816
- [Background] Beal DS, Quraan MA, Cheyne DO, Taylor MJ, Gracco VL, De Nil LF. Speech-induced suppression of evoked auditory fields in children who stutter. Neuroimage. 2011 Feb 14;54(4):2994-3003. doi: 10.1016/j.neuroimage.2010.11.026. Epub 2010 Nov 21. PMID 21095231
- [Background] Beal DS, Cheyne DO, Gracco VL, Quraan MA, Taylor MJ, De Nil LF. Auditory evoked fields to vocalization during passive listening and active generation in adults who stutter. Neuroimage. 2010 Oct 1;52(4):1645-53. doi: 10.1016/j.neuroimage.2010.04.277. Epub 2010 May 7. PMID 20452437
- [Background] Daliri A, Max L. Stuttering adults' lack of pre-speech auditory modulation normalizes when speaking with delayed auditory feedback. Cortex. 2018 Feb;99:55-68. doi: 10.1016/j.cortex.2017.10.019. Epub 2017 Nov 13. PMID 29169049
- [Background] Daliri A, Max L. Modulation of auditory processing during speech movement planning is limited in adults who stutter. Brain Lang. 2015 Apr;143:59-68. doi: 10.1016/j.bandl.2015.03.002. Epub 2015 Mar 18. PMID 25796060
- [Background] Daliri A, Max L. Electrophysiological evidence for a general auditory prediction deficit in adults who stutter. Brain Lang. 2015 Nov;150:37-44. doi: 10.1016/j.bandl.2015.08.008. Epub 2015 Aug 31. PMID 26335995
- [Background] Park CH, Park TW, Yang JC, Lee KH, Huang GB, Tong Z, Park MS, Chung YC. No negative symptoms in healthy volunteers after single doses of amisulpride, aripiprazole, and haloperidol: a double-blind placebo-controlled trial. Int Clin Psychopharmacol. 2012 Mar;27(2):114-20. doi: 10.1097/YIC.0b013e3283502773. PMID 22241281
- [Background] Tran NL, Maguire GA, Franklin DL, Riley GD. Case report of aripiprazole for persistent developmental stuttering. J Clin Psychopharmacol. 2008 Aug;28(4):470-2. doi: 10.1097/JCP.0b013e31817ea9ad. No abstract available. PMID 18626285
- [Background] Kim BU, Kim HW, Park EJ, Kim JH, Boon-Yasidhi V, Tarugsa J, Reyes A, Manalo SG, Joung YS. Long-Term Improvement and Safety of Aripiprazole for Irritability and Adaptive Function in Asian Children and Adolescents with Autistic Disorder: A 52-Week, Multinational, Multicenter, Open-Label Study. J Child Adolesc Psychopharmacol. 2022 Sep;32(7):390-399. doi: 10.1089/cap.2022.0004. PMID 36112116
- [Background] Maguire GA, Nguyen DL, Simonson KC, Kurz TL. The Pharmacologic Treatment of Stuttering and Its Neuropharmacologic Basis. Front Neurosci. 2020 Mar 27;14:158. doi: 10.3389/fnins.2020.00158. eCollection 2020. PMID 32292321
- [Background] Alm PA. The Dopamine System and Automatization of Movement Sequences: A Review With Relevance for Speech and Stuttering. Front Hum Neurosci. 2021 Dec 2;15:661880. doi: 10.3389/fnhum.2021.661880. eCollection 2021. PMID 34924974